CLINICAL TRIAL: NCT02723981
Title: Prospective, Multi-centre, Randomized, Parallel Comparison to Evaluate the Safety and Efficacy of the Abluminal Sirolimus Coated Bio-engineered Stent (COMBO Stent) in Association With Short-term Single Antiplatelet Therapy in Patients With Coronary Artery Disease With an Indication for Chronic Oral Anticoagulant Therapy as Compared to a Guidelines-based Strategy
Brief Title: COMBO-Stent in Patients on Chronic Anticoagulant Therapy (COSTA) COSTA-Bleed and COSTA-Outcome Trials
Acronym: COSTA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Regulatory authority approval for the initial study design could not be obtained
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: OrbusNeich (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COSTA-MPG-001
Record Dates: First submitted 2016-03-16; First posted 2016-03-31 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Stable Angina; Unstable Angina; STEMI; NSTEMI; Coronary Disease
Keywords: Stent , COMBO Stent, anticoagulation
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Disease | interventions — Clopidogrel; Rivaroxaban; Dabigatran; Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COMBO-Stent (Experimental): Implantation of COMBO-Stent and medication with (N)OAC and clopidogrel for 3 months followed by (N)OAC alone
  Interventions: Device: COMBO-Stent; Drug: Clopidogrel, Vitamin K Antagonist, Rivaroxaban, Dabigatran
- Any Drug eluting or bare metal stent (Active Comparator): Implantation of any drug eluting oder bare metal stent combined with anticoagulant medication according to ESC guidelines
  Interventions: Device: Any drug eluting stent oder bare metal sent; Drug: ASA, Clopidogrel, Vitamin K Antagonist, Rivaroxaban, Dabigatran

INTERVENTIONS:
Device: COMBO-Stent — The OrbusNeich COMBO Bio-engineered Sirolimus Eluting Stent (COMBO Stent) consists of a 316L stainless steel alloy abluminally coated with a biocompatible, biodegradable poly-mer containing sirolimus. Covalently attached to the surface of the stent is a layer of murine, monoclonal, anti-human CD34 antibody. The antibody specifically targets circulatory CD34+ cells (endothelial progenitor cells) thus favoring endothelialization.
  Arms: COMBO-Stent
Drug: Clopidogrel, Vitamin K Antagonist, Rivaroxaban, Dabigatran — Anticoagulant medication after stent Implantation: (N)OAC and clopidogrel for 3 months followed by (N)OAC
  Other Names: Plavix, Marcumar, Xarelto, Pradaxa
  Arms: COMBO-Stent
Device: Any drug eluting stent oder bare metal sent — Implantation of traditional bare metal stents and/or drug eluting stents (any device approved on the market, implanted according to CE marking and IFU) and medication regimen in accordance with ESC Guidelines
  Other Names: Cypher, Taxus, CoStar, Janus, Endeavor, Xience, Promus, Multi Link, Coroflex, Veriflex, Integrity, Driver
  Arms: Any Drug eluting or bare metal stent
Drug: ASA, Clopidogrel, Vitamin K Antagonist, Rivaroxaban, Dabigatran — A combination of antiplatelet and anticoagulant therapy according to ESC guidelines (2014)
  Other Names: Anticoagulant medication according to ESC guidelines
  Arms: Any Drug eluting or bare metal stent

SUMMARY:
Prospective, multi-centre, randomized, open-label, parallel comparisons to evaluate

* the incidence of bleedings (COSTA-Bleed) and
* the incidence of ischemic and bleeding events (COSTA-Outcome) following a therapy with the abluminal sirolimus coated bio-engineered stent (COMBO stent) in association with short-term single antiplatelet therapy as compared to a guidelines-based strategy in patients with coronary artery disease with an indication for chronic oral anticoagulant therapy.

DETAILED DESCRIPTION:
The COSTA trials are investigator-initiated studies aimed at comparing the clinical outcome after percutaneous coronary intervention (PCI) using a COMBO-stent based strategy associated with short-term antiplatelet therapy with a guidelines-based therapy in patients with an indication for chronic oral anticoagulation. The study is organized as a national, multi-centre prospective, randomized trial. The duration of the follow-up is 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older;
* Willingness to comply with the study protocol; subject or a legally authorized representative must provide written informed consent prior to any study related procedure, in accordance with International Conference on harmonization of Good Clinical Practice (ICH-GCP) guidelines and per site requirements.
* Patients on anticoagulant therapy or treatment-naive pa-tients with an indication to chronic anticoagulant therapy. Indications to oral anticoagulation may include atrial fibrillation, prosthetic valve disease, peripheral by-pass surgery, lung embolism or deep vein thrombosis or any other indication according to the Investigator´s opinion.
* Single or multiple de novo lesion in a native coronary artery, all amenable to treatment with the COMBO stent;

Exclusion Criteria:

* Patients who, in the Investigator's opinion, should not be treated with (N)OAC. These may include, for instance: history of BARC 3-5 bleeding <12 months; patients with a haemorrhagic disorder or bleeding diathesis (e.g. von Willebrand disease, haemophilia A or B or other hereditary bleeding disorder, history of spontaneous intra-articular bleeding, history of prolonged bleeding after surgery/intervention); patients with recent major surgery; history of intraocular, spinal, retroperitoneal, intra-articular or recent gastrointestinal bleeding unless the causative factor has been permanently eliminated or repaired; (reduction in the haemoglobin level of at least 2g/dL, transfusion of at least two units of blood, or symptomatic bleeding in a critical area or organ) including life-threatening bleeding episode (symptomatic intracranial bleeding, bleeding with a decrease in the haemoglobin level of at least 5g/dL or bleeding requiring transfusion of at least 4 units of blood or inotropic agents or necessitating surgery); Anaemia (haemoglobin <10g/dL) or thrombocytopenia including heparin-induced thrombocytopenia (platelet count <100E9/L) at screening;
* Pregnant or nursing patients. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test;
* Other medical illness with a life expectancy <2 years (e.g. known malignancy) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol or confound the data in-terpretation or is associated with a limited life expectancy;
* Patient has received an organ transplant or is on a wait-ing list for an organ transplant;
* Known hypersensitivity or contraindication to antiplate-let or anticoagulant agents that does not allow guide-lines-compliant therapy and that cannot be adequately pre-medicated;
* Previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti-Murine Antibodies (HAMA);
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Current participation in another investigational drug or device study except for non-interventional registries;
* Patients not willing or able to comply with the protocol requirements or considered unreliable by the Investigator concerning the requirements for follow up during the study and/or compliance with study drug administration;

Angiographic exclusion criteria:

* Vessel diameter <2 und > 5mm;
* Target lesion with characteristics that make it unsuitable for stent delivery and deployment;
* Planned use of a stent or another coronary device in the same or another session (target vessel or non-target vessel), precluding a COMBO-only strategy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with bleedings | 6 weeks
  any BARC (bleeding academic research consortium) bleeding at 6 weeks - superiority.
Number of patients with safety events | 15 months
  Strategy oriented composite safety endpoint, including death (unless proven not to be connected to the other endpoints), any MI, stroke or systemic embolism, definite or probable stent thrombosis, BARC 3-4 bleeding at 15 months post PCI - non-inferiority with reflex to superiority testing. Hierarchical testing: Endpoint II is only tested if null hypothesis of no difference in bleeding incidence can be rejected at final analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tommasso Gori, Principal Investigator — Universitaetsmedizin Mainz; Ibrahim Akin, Principal Investigator — Universitaetsmedizin Mannheim
Locations (10):
- Germany (10):
  - MVZ am Kuechwald GmbH, Chemnitz
  - Elisabeth Krankenhaus, Essen
  - Universitaetsmedizin Mainz, Mainz
  - Theresienkrankenhaus und St. Hedwig GmbH, Mannheim
  - Universitaetsmedizin Mannheim, Mannheim
  - St. Franziskus, Kliniken Maria Hilf GmbH, Mönchengladbach
  - Evangelisches Krankenhuas Muehlheim a.d. Ruhr GmbH, Muehlheim An Der Ruhr
  - Diakonissen-Stiftungs-Krankenhaus, Speyer
  - Herzklinik Ulm GbR, Ulm
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No